CLINICAL TRIAL: NCT06327711
Title: Proof of Concept Study: Long-term Benefits of a Blend of Nutritional Ingredients for Type 2 Diabetes
Brief Title: Benefits of Nutritional Ingredients for Type 2 Diabetes
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Change in study scope
Sponsor: Abbott Nutrition (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: BL77
Record Dates: First submitted 2024-02-07; First posted 2024-03-25 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-12

CONDITIONS: Diabetes type2

STUDY DESIGN:
Intervention Model Description: 2 groups, non-crossover
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CHO Blend (Active Comparator): Group will consume a ready to feed CHO blend beverage
  Interventions: Other: Control: CHO Blend
- CHO Blend plus AN100 (Experimental): Group will consume a ready to feed CHO plus AN100 beverage
  Interventions: Other: Experimental: CHO Blend plus AN100

INTERVENTIONS:
Other: Control: CHO Blend — 2 servings as a snack or between meals morning and evening
  Arms: CHO Blend
Other: Experimental: CHO Blend plus AN100 — 2 servings as a snack or between meals morning and evening
  Arms: CHO Blend plus AN100

SUMMARY:
This is a prospective randomized, double-blinded, parallel design study to evaluate the benefits of long-term consumption of two experimental blends of liquid supplements.

ELIGIBILITY:
Inclusion Criteria:

* Has type 2 diabetes
* Taking a maximum of 3 oral anti-diabetic drugs, one must be Metformin.
* HbA1c ≥ 6.5% and ≤ 9.5% based on blood sample obtained at Screening Visit
* BMI > 27.0 and < 35.0 kg/m2
* Weight is stable for the two months prior to Baseline visit
* Either male or a non-pregnant, non-lactating female, at least 6 weeks postpartum prior to Baseline Visit
* If on chronic medication type and dose were constant for at least two months prior to the baseline Visit, and medication will continue throughout the study
* Willingness to follow the protocol as described, including consumption of study product and completing any forms/questionnaires needed throughout the study
* Four-week washout period between completion of a previous research study that required ingestion of any study food or drug and start in current study
* The participant is willing to refrain from taking non-study diabetes-specific oral nutritional formulas during the study

Exclusion Criteria:

* Use of exogenous insulin or GLP1 agonists
* Follows a non-typical eating pattern such as very low carbohydrate diet
* Pregnant or attempting to conceive
* Confirmed type 1 diabetes and/or history of diabetic ketoacidosis
* Current infection inpatient surgery or received systemic corticosteroid treatment in last 3 months; or received antibiotics in last 3 weeks
* Has current active malignant disease or treated within the last 6 months for cancer, except basal or squamous cell skin carcinoma
* Significant cardiovascular event within 6 months prior or history of congestive heart failure
* End-stage organ failure or is post-organ transplant
* Current or history of renal disease, on dialysis or severe gastroparesis
* Diagnosed hepatic disease or late stage liver fibrosis. Participants with prevalent angina will not be excluded.
* Had bariatric surgery including gastric balloon; history of gastrointestinal disease or intestinal surgery
* Chronic, contagious, infectious disease
* Eating disorder, severe dementia or delirium, history of significant neurological or psychiatric disorder, alcoholism, substance abuse or any other conditions that may interfere with study product consumption or compliance with study protocol procedures
* Taking any herbals, dietary supplements, or medications during the past four weeks prior to baseline visit that could profoundly affect blood glucose, body weight, muscle, metabolism, appetite or microbiome incretin mimetics, other drugs indicated for weight loss, cannabis, glucocorticoids, probiotic supplements). Those who have stopped using such supplements/ medications for ≥4 weeks prior to baseline need not be excluded).
* Using diabetes-specific oral nutritional supplements(s), defined as more than one eating occasion per week within the past 4 weeks (those users who can stop using such products for ≥4 weeks before baseline visit need not be excluded)
* Actively enrolled in a weight loss program
* Clotting or bleeding disorders
* Blood or blood-related diseases
* Blood transfusion within the last 3 weeks
* Allergic or intolerant to any ingredient found in the study products
* Engages in strenuous exercise duration of 1 hour or longer, 3 or more times per week
* Participates in another study that has not been approved as a concomitant study by Abbott Nutrition
* Participant has skin lesions hyperhidrosis, eczema, psoriasis, scarring, tattoos, redness, infection or edema at the application sites that could interfere with device placement or accuracy of interstitial glucose measurements

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-09 (Estimated); Primary Completion 2025-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Matsuda Index | Baseline to week 12
  Change in insulin sensitivity
Fasted Glucose | Baseline week 4, week 8 and week 12
  Change in fasted glucose levels overtime
Fasted Insulin | Baseline week 4, week 8 and week 12
  Change in fasted insulin levels overtime

SECONDARY OUTCOMES:
Body Weight | Baseline up to 12 weeks
  Changes in body weight
Body Composition Measurements | Baseline up to 12 weeks
  Changes in bio electrical impendence analysis (BIA)
Continuous Glucose Monitoring | Baseline, week 1 to week 2, week 11 and 12
  Change in glycemic variability
Glycated Hemoglobin | Baseline week 4, week 8 and week 12
  Change in hemoglobin A1c
Resting Energy Expenditure (REE) | Baseline to week 12
  Changes in REE
Microbiome - Fecal | Baseline week 2, week 4, week 8 and week 12
  Changes in fecal microbiome
Microbiome - Saliva | Baseline week 2, week 4, week 8 and week 12
  Changes in saliva microbiome
Waist Circumference | Baseline up to 12 weeks
  Changes in waist circumference
Hip Circumference | Baseline up to 12 weeks
  Changes in hip circumstance
Conicity Index | Baseline up to 12 weeks
  Changes in conicity index

OTHER OUTCOMES:
Blood Pressure | Baseline week 4, week 8 and week 12
  Systolic and Diastolic
Accelerometry Data | Baseline to week 12
  Change in accelerometer daily activities
Diabetes Distress Scale | Baseline to week 12
  Participant assessed 29 questions rated from 1 to 5 were higher number if less favorable
Dietary Intake | Baseline to week 12
  Energy and macronutrient intake calculated from participant reported diary
Blood biomarkers - inflammation | Time Frame: Baseline to week 12
  Change in protein marker of inflammation such as CRP
Urine biomarkers - inflammation | Time Frame: Baseline to week 12
  Change in protein marker of inflammation such as CRP

CONTACTS AND LOCATIONS:
Overall Officials: Suzette Pereira, Study Chair — Abbott Nutrition
Locations (1):
- Kent State University, Kent, Ohio, United States